CLINICAL TRIAL: NCT07240870
Title: Age-dependent EEG Coupling, Periodic and Aperiodic Characteristics During Desflurane Anesthesia From Adults to Elderlies
Brief Title: Age-dependent EEG Characteristics During Desflurane Anesthesia From Adults to Elderlies
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director, Chinese PLA General Hospital
Other Study IDs: PLAGH-Des-EEG
Record Dates: First submitted 2025-09-29; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: EEG; Aging; Desflurane Anesthesia
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18-40 years age group: 18-40 years
  Interventions: Other: Age
- 40-65 years age group: 40-65 years
  Interventions: Other: Age
- >65 years age group: >65 years
  Interventions: Other: Age

INTERVENTIONS:
Other: Age — Divided into three age groups based on the age of the included patients

SUMMARY:
This study is a prospective cohort study that records bilateral frontal EEG data from patients undergoing elective non-cardiac or non-neurosurgical surgeries and divides them into different age groups based on age. All patients received maintenance of general anesthesia with desflurane, and the periodic and aperiodic components, permutation cross mutual information (PCMI), and phase lag entropy (PLE) of EEG data were analyzed under different states of wakefulness, general anesthesia, and recovery. Professional correlation analysis methods were used to analyze the EEG spectrum.

DETAILED DESCRIPTION:
This study investigates how the aging brain responds to general anesthesia (GA). As global populations grow older, an increasing number of elderly patients require surgery with GA. However, the aging brain undergoes significant changes, such as a reduction in brain volume (atrophy) and a decreased ability to metabolize drugs. These factors can make anesthesia riskier for older adults, potentially leading to complications like delayed recovery or post-operative cognitive dysfunction. Currently, most anesthesia monitoring systems are designed based on data from younger, healthier adults and may not accurately reflect the brain state of an elderly patient. This study aims to address this critical gap by analyzing the brain's electrical signals (via EEG) across different age groups to understand how aging influences the brain's response to anesthesia.

The research team enrolled 47 patients, aged between 19 and 82 years, who were scheduled for surgery requiring general anesthesia with desflurane. Participants were divided into three age groups for comparison: young adults (18-40 years), middle-aged adults (40-65 years), and older adults (over 65 years). The investigators analyzed the periodic and aperiodic component, permutation cross mutual information (PCMI) and phase lag entropy (PLE) of EEG data in the states of awake, GA, and recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female not limited
2. Patients who undergo elective non cardiac surgery or non neurosurgical surgery;
3. ASA classification levels 1-3

Exclusion Criteria:

1. Individuals with central nervous system disorders such as autism, attention deficit/hyperactivity disorder, epilepsy, or any congenital mental illness;
2. Patients with any contraindications to the use of desflurane, such as those with a history of malignant hyperthermia (MH), allergies to halogenated anesthetics, and patients with significantly elevated intracranial pressure (ICP);
3. Patients with unstable clinical conditions, such as severe hypotension or circulatory failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram-derived Features | Assessed from 2-minute EEG segments at each of three states: Baseline, Under General Anesthesia, and Recovery.
  The following quantitative features will be extracted and assessed from the electroencephalogram (EEG) recordings:
  Periodic Component: The oscillatory power within standard frequency bands: Delta (1-4 Hz), Theta (4-8 Hz), Alpha (8-13 Hz), Beta (13-30 Hz), and Gamma (30-45 Hz).
  Aperiodic Component: The offset and exponent of the background '1/f' activity, extracted via spectral parameterization.
  Permutation Cross Mutual Information (PCMI): A measure to assess nonlinear coupling and directional information flow between different brain regions.
  Phase Lag Entropy (PLE): A measure to evaluate the dynamic stability of functional brain connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- First Medical center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No